CLINICAL TRIAL: NCT05664139
Title: A Prospective, Single-arm Study on the Efficacy and Safety of Recombinant Human Adenovirus Type 5 Injection Combined With PD-1 Monoclonal Antibody and Nab-paclitaxel in the Treatment of Patients With Liver Metastases From Malignant Melanoma
Brief Title: Recombinant Human Adenovirus Type 5 Injection Combined With PD-1 Monoclonal Antibody and Nab-paclitaxel in the Treatment of Patients With Liver Metastases From Malignant Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry); SunWay Biotech Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJCH-HR-001
Record Dates: First submitted 2022-12-08; First posted 2022-12-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Malignant Melanoma; Liver Metastases
Keywords: recombinant human adenovirus type 5; Camrelizumab; Nab-paclitaxel; Malignant Melanoma; Liver Metastases
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): * Recombinant Human Adenovirus Type 5 Injection: 1ml or 2ml, d1, q3w, 4 cycles;
  * Camrelizumab: 200mg, d2, q3w;
  * Nab-paclitaxel: 260mg/m2, d1, q3w, 4-6 cycles;
  Interventions: Drug: Recombinant Human Adenovirus Type 5 Injection,Camrelizumab,Nab-paclitaxel

INTERVENTIONS:
Drug: Recombinant Human Adenovirus Type 5 Injection,Camrelizumab,Nab-paclitaxel — Recombinant Human Adenovirus Type 5 Injection:①the longest diameter of the lesion≥10mm and≤40mm, inject 1ml into the tumor each time;②the longest diameter of the lesion≥40mm and≤80mm, inject 2ml into the tumor each time. planned injections at D1. Every 3 weeks is a period, a total of 4 cycles; if there are visceral and superficial lesions at the same time, the injection lesions will be selected by the investigator based on possible benefits.
  Camrelizumab:200mg/time.Intravenous within 48 hours after injection of recombinant human adenovirus type 5 injection. Every 3 weeks is a period, and the treatment is continued until the subject has disease progression or unacceptable toxicity or death.
  Nab-paclitaxel:260mg/m2, D1, every 3 weeks as a period, a total of 4-6 cycles (determined by the investigator), or continue treatment until the subject has disease progression or Intolerable toxicity or death.

SUMMARY:
This study is the first to explore the efficacy and safety of recombinant human adenovirus type 5 injection combined with PD-1 monoclonal antibody and nab-paclitaxel in the treatment of patients with liver metastases of melanoma, in order to provide a new method for the clinical treatment of melanoma. The model also provides reference and basis for other tumor treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, and ≤ 75 years old, gender is not limited;
2. Patients with liver metastasis of malignant melanoma diagnosed by histopathology;
3. There must be an injectable lesion in the liver, and the lesion must meet the requirements of RECIST 1.1 measurable target lesion;
4. The liver lesion needs to be judged by the surgeon to have a poor prognosis in biological behavior; or the surgeon judges that it can be resected, but the patient refuses the operation, and the liver metastases must meet the following requirements:

   1. The number of metastatic lesions should not exceed 5, and the sum of the longest diameters of the total metastatic lesions must be ≤100mm;
   2. The longest diameter of a single lesion ≤ 100 mm;
   3. The longest diameter of the injection lesion must be ≥10mm and ≤80mm;
5. ECOG physical condition score 0-1 points;
6. Expected survival time > 3 months;
7. Laboratory examinations meet the following standards:

   1. White blood cell count ≥3.0×109/L, absolute value of neutrophils ≥3.0×109/L, platelet count ≥100×109/L, hemoglobin ≥90g/L;
   2. International normalized ratio (INR) ≤ 1.5, and activated partial thromboplastin time (APTT) ≤ 1.5 × upper limit of normal (ULN) or partial prothrombin time (PTT) ≤ 1.5 × ULN;
   3. Total bilirubin ≤ 1.5×ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN;
   4. Serum creatinine ≤1.5×ULN or creatinine clearance ≥50ml/min at 24 hours.
8. The interval between the date of the first treatment in this study and the date of the last anti-tumor treatment in the past is ≥14 days, and the adverse reactions of the previous anti-tumor treatment have recovered to baseline or below grade 1 [evaluation criteria for common adverse events (CTCAE version 5.0)] (hair loss and grade 2 anemia);
9. Volunteer to participate in this study and sign the informed consent;
10. Female patients of childbearing age or male patients whose sexual partner is female of childbearing age should take effective contraceptive measures throughout the treatment period and 6 months after the last medication.

Exclusion Criteria:

1. Bone metastasis, lymph node metastasis, brain metastasis and other metastatic malignant melanoma;
2. njectable lesions have previously received other local treatments such as ablation, intervention, and Haifu Knife;
3. Patients who have previously received oncolytic virus drugs (such as T-VEC) or other similar drugs;
4. Patients who have previously received PD-1/PD-L1/PD-L2 therapy;
5. Local lesions cannot meet the volume requirements for intratumoral injection or are not suitable for intratumoral injection;
6. Accompanied by malignant pleural effusion and ascites;
7. Patients who are positive for hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) antibody;
8. People who are known to be allergic to the study drug or its active ingredients, or have a history of allergy to similar biological agents;
9. Received antiviral drug treatment within 4 weeks before enrollment, such as acyclovir, ganciclovir, valaciclovir, vidarabine, etc.;
10. Received any other experimental drugs or participated in other interventional clinical trials within 4 weeks before enrollment;
11. Pregnant or lactating women, men or women who are unwilling to take effective contraceptive measures;
12. Vulnerable groups: including the mentally ill, critically ill subjects, minors, cognitively impaired, etc.;
13. Child-Pugh C Evidence of liver function or hepatocyte decompensation, including refractory ascites, bleeding from esophageal or gastric varices, and hepatic encephalopathy;
14. There is a history of immunodeficiency or autoimmune disease, or receiving long-term systemic steroid therapy or any form of immunosuppressive therapy within 7 days before enrollment;
15. Patients with a history of active tuberculosis (TB), active hepatitis, patients who have been evaluated for oral nucleoside (acid) analogues, known human immunodeficiency virus (HIV) positive patients, other serious infections that require treatment, and those who are taking anti-inflammatory drugs Viral drugs or large doses of adrenal corticosteroids;
16. Accompanied by any unstable systemic diseases, including but not limited to: hypertensive patients whose blood pressure cannot be lowered to normal, uncontrolled diabetes, cerebrovascular accident or transient cerebral ischemia, mental abnormality or active cerebral hemorrhage, not Stable angina, myocardial infarction (a history of myocardial infarction of 6 months or more is allowed), congestive heart failure, severe arrhythmia requiring drug therapy, severe cardiopulmonary disease abnormality, renal or metabolic disease, severe liver dysfunction ( including severe jaundice, hepatic encephalopathy, refractory ascites, or hepatorenal syndrome);
17. Having other malignant tumors in the past or at the same time, except for the following: stage I uterine cancer that has been radically cured, localized prostate cancer that is currently considered cured after radical surgery, and other solid tumors that have been cured for more than 5 years and have no signs of recurrence;
18. Known central nervous system tumors, including metastatic brain tumors;
19. Combined with medical contraindications that cannot accept any contrast-enhanced imaging examination (CT or MRI);
20. The investigator judges that the patient has other conditions that are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response rate (ORR) | 1 year
  From the first administration of the study drug to disease progression, unacceptable toxicity, withdrawal of informed consent or termination of the study (up to 1 year), including the proportion of CR and PR among all patients.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 1 year
  It refers to the proportion of patients whose tumor shrinks or stabilizes and keeps for a certain period of time, including CR, PR and SD cases among all patients.
Progression-free survival (PFS) | 1 year
  The time (days) from the date of randomization to the first observation of disease progression (based on imaging), if the patient died of other causes before disease progression, the time from the date of randomization to death was calculated number of days.
One-year Overall Survival | 1 year
  1-year overall survival rate
Quality of life (QoL) | 1 year
  EORTC QLQ-C30
Adverse event collection | 1 year
  Incidence of adverse reactions

OTHER OUTCOMES:
Pathological changes of injection lesions | 1 year
  Detection of pathologically-based changes in injected lesions
MRI-based changes in injected lesions | 1 year
  Detection of MRI-based changes in injected lesions
Changes of CD4+ cells count, CD8+ cells count, Th1 cells count, Th2 cells count, Treg cells count in peripheral blood | 1 year
  Changes of CD4+ cells count, CD8+ cells count, Th1 cells count, Th2 cells count, Treg cells count in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chen, PhD, Study Director — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: No